CLINICAL TRIAL: NCT02519673
Title: Comparison of Corneal Stromal Tissue Consumption Values Estimated When Programming the Intervention Versus the Values Measured by Pre and Postoperative Topography
Brief Title: Comparison of Corneal Stromal Tissue Consumption (LATAC)
Acronym: LATAC
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: JFO_2015_26
Record Dates: First submitted 2015-08-04; First posted 2015-08-11 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Disorders, Refractive
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Measurement of stromal tissue ablation — Stromal tissue consumption will be estimated preoperatively by WaveLight Allegretto EX-500 laser and central corneal thickness will be measured by Pentacam. One month after refractive surgery, during follow-up,central corneal thickness will be again measured by Pentacam.

SUMMARY:
In refractive surgery, stromal ablation depth is fundamental because it determines the thickness of the residual posterior wall. The posterior wall is an essential element that guarantees the refractive stability and the long term prevention of corneal ectasia after corneal refractive surgery. A minimum thickness of more or less 300 microns is universally accepted. Its calculation is based on well-known formulas, such as Munnerlynn ones.

With the excimer laser platform last generation WaveLight® Allegretto® EX-500 of Alcon, a new treatment option called "wavefront optimized" is offered for myopia, astigmatism and hyperopia. The ablation profile has been developed to save stromal tissue consumption and to favor the quality of vision, by optimizing connections between the optical zone and the transition zone of the photoablation. Alongside the theoretical formulas, evaluation of the depth of ablation may be defined by differential ultrasonic pachymetry or by topographical analysis pre and postoperatively. The latter is currently the method of reference to assess the corneal thickness.

ELIGIBILITY:
Inclusion Criteria:

* Patients having a refractive disorder and for whom a refractive surgery is programmed.

Exclusion Criteria:

* Patient opposed to participation in the study
* Another refractive surgery technique
* Hyperopic patient
* Pregnant or lactating woman
* Patient under a measure of legal protection
* Absence of affiliation to social security or universal health coverage (CMU)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having a refractive disorder and for whom a refractive surgery by LASIK is programmed.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-08-08 (Actual); Primary Completion 2017-01-18 (Actual); Study Completion 2017-03-15 (Actual)

PRIMARY OUTCOMES:
Difference between stromal tissue consumption, expressed in micrometers, estimated before surgery by WaveLight Allegretto EX-500 laser and measured one month after surgery by Pentacam | One month
  Stromal tissue consumption will be estimated preoperatively by WaveLight Allegretto EX-500 laser and central corneal thickness will be measured by Pentacam. One month after refractive surgery, during follow-up,central corneal thickness will be again measured by Pentacam. The difference between the estimated and the measured tissue consumption will be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation ophtalmique Adolphe de Rothschild, Paris, Paris, France